CLINICAL TRIAL: NCT01419886
Title: Testing of a New Scale Measuring Medical Outcomes of Dysphagia (MOD) in Adult Patients With Swallowing Disorders
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Other Study IDs: CIHR-93685, CCSRI-020190
Record Dates: First submitted 2011-08-04; First posted 2011-08-18 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dysphagia

SUMMARY:
Swallowing disorders (dysphagia) are common in adult patients. There is emerging evidence that dysphagia itself can cause adverse medical outcomes. There is a three-fold increased risk for pneumonia in these patients versus similar patients without dysphagia. Patients with dysphagia also suffer poor nutrition and dehydration. Patients can become so malnourished that it slows their recovery. Dysphagia can cause choking when food or liquid enters the lungs. Over time, this will cause pneumonia and even death. More acutely, patients fear that their choking will cause them to suffocate and die. Over time, patients are embarrassed to be seen choking and thus feel forced to dine alone. These patients report feelings of isolation and depression. To date, there are no practical methods to assess these adverse outcomes of swallowing difficulties in patients. This research will be the first to address this gap. Specifically, as part of previous research (PhD dissertation by RM, the PI) a new measure of medical outcomes of dysphagia was developed, titled the Medical Outcomes of Dysphagia (MOD) scale. The MOD consists of 3 subscales that each measure lung, nutrition-hydration or psychological consequences in patients with swallowing difficulties. Unlike more expensive and complex tests, the MOD has been designed for both in- and outpatients. This research will validate each MOD subscale to ensure retention of only items that are reliable and valid for use with patients who have dysphagia due to any disease etiology. The final MOD subscales will be the first to allow clinicians to track medical complications in their patients and to ensure that treatment is effective. Globally, the MOD subscales will direct limited health care resources to the most effective treatments for swallowing disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years)
* Any disease etiology, including but not limited to: previous or current diagnosis of head and neck cancer (treatment may include surgery, radiation or chemotherapy, or a combination of more than one), stroke, cervical spine abnormality, brain tumour, cardiovascular surgery, and Parkinson's disease
* Current diagnosis of dysphagia, as determined by a speech language pathologist
* English-speaking

Exclusion Criteria:

* No dysphagia
* Cognitive impairment
* Limited fluency in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients of the University Health Network who have a diagnosis of dysphagia.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2010-10; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Reliability of the MOD subscales | 24 hours
  Inter-rater reliability will be assessed using the Intraclass Correlation Coefficient (ICC). The MOD is being standardized for clinical purposes; therefore sufficient reliability will be set high at an ICC>0.90
Validity of the MOD subscales | 24 hours
  Rasch analysis will be used to: i) develop three separate interval-level MOD subscales each with items mapped along a linear continuum of impairment severity; ii) identify and eliminate redundant items within each subscale, allowing for shorter MOD subscales with less respondent burden, and iii) ensure item properties within each subscale are invariant so that the MOD subscales will work well with a variety of patients regardless of disease type.

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Martino, PhD, Principal Investigator — University of Toronto / University Health Network
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Martino R, Beaton D, Diamant NE. Perceptions of psychological issues related to dysphagia differ in acute and chronic patients. Dysphagia. 2010 Mar;25(1):26-34. doi: 10.1007/s00455-009-9225-0. Epub 2009 Aug 6. PMID 19657695
- [Background] Martino R, Beaton D, Diamant NE. Using different perspectives to generate items for a new scale measuring medical outcomes of dysphagia (MOD). J Clin Epidemiol. 2009 May;62(5):518-26. doi: 10.1016/j.jclinepi.2008.05.007. Epub 2008 Aug 22. PMID 18722085
- See also: Related Info — http://swallowinglab.uhnres.utoronto.ca/